CLINICAL TRIAL: NCT05665374
Title: General Use-Results Study of Calquence Capsules 100 mg in Patients With Previously Untreated Chronic Lymphocytic Leukaemia (Including Small Lymphocytic Lymphoma)
Brief Title: Calquence CLL 1L Japan PMS _ Japan Post-Marketing Surveillance (PMS) Study
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D822EC00001
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Previously Untreated Chronic Lymphocytic Leukaemia (Including Small Lymphocytic Lymphoma)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
To understand the incidence of ADRs of Calquence capsules 100 mg (acalabrutinib) used in patients with previously untreated chronic lymphocytic leukaemia (CLL) (including small lymphocytic lymphoma (SLL)) in the post-marketing setting under actual use

DETAILED DESCRIPTION:
To understand the incidence of ADRs of Calquence capsules 100 mg (acalabrutinib) (hereinafter referred to as "CALQUENCE") used in patients with previously untreated chronic lymphocytic leukaemia (CLL) (including small lymphocytic lymphoma (SLL)) in the post-marketing setting under actual use.

This investigation will be conducted as the additional pharmacovigilance activity specified in the Japan Risk Management Plan (J-RMP) of CALQUENCE, in compliance with the Ministerial Ordinance on Good Post-marketing Study Practice (GPSP Ordinance) and for the purpose of application for re-examination under Article 14-4 of the Law for Ensuring Quality, Efficacy, and Safety of Drugs and Medical Devices (PMD Act).

ELIGIBILITY:
Inclusion Criteria:

Patients with previously untreated chronic lymphocytic leukaemia (including small lymphocytic lymphoma) who are treated with Calquence for the first time will be enrolled in the study after the approval date of the sJNDA for the additional indication.

-

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with previously untreated chronic lymphocytic leukaemia (including small lymphocytic lymphoma) who are treated with Calquence
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADRs | 24 weeks
  the incidence of ADRs related to Calquence Safety Specifications : infection, bone marrow depression

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (15):
- Japan (15):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hyōgo
  - Research Site, Kanagawa
  - Research Site, Kyoto
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nara
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home